CLINICAL TRIAL: NCT03665883
Title: Randomised Controlled Trial on Use of Monopolar Energy Versus Blunt Dissection in Totally Extra-peritoneal Hernioplasty (TEP) for Inguinal Hernia - the Effect on the Output of Pre-peritoneal Drain
Brief Title: Use of Diathermy Versus Blunt Dissection in TEP for Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Joe King-Man Fan, Honorary Consultant, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HERN-MONOPOLAR-01
Record Dates: First submitted 2018-08-31; First posted 2018-09-11 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Seroma; Hernia, Inguinal
MeSH Terms: conditions — Seroma; Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: the effect on seroma formation and output of pre-peritoneal drain after TEP by monoploar diathermy or blunt dissection approach will be studied
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, assessors and investigators will be blinded on patient group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diathermy preferred (Active Comparator): Monopolar energy is the preferred dissection approach in this group of patients undergo TEP. Total time of activation of monopolar machine will recorded by specially designed device
  Interventions: Procedure: Monopolar energy
- Blunt dissection preferred (Active Comparator): Blunt dissection is the preferred dissection approach in this group of patients undergo TEP. Use of monopolar energy for haemostasis is still allowed upon surgeons' decision. Total time of activation of monopolar machine will recorded by specially designed device
  Interventions: Procedure: Blunt dissection

INTERVENTIONS:
Procedure: Monopolar energy — Monopolar energy in TEP for inguinal hernia
  Arms: Diathermy preferred
Procedure: Blunt dissection — Blunt dissection in TEP for inguinal hernia
  Arms: Blunt dissection preferred

SUMMARY:
There is a long debate whether monopoloar or blunt dissection should be adopted in TEP to minimise the chance of seroma formation. This study aims at study the effect on seroma formation (and pre-peritoneal drain output) by 2 techniques in randomised controlled trial.

DETAILED DESCRIPTION:
There is a long debate whether monopoloar or blunt dissection should be adopted in TEP to minimise the chance of seroma formation. This study aims at study the effect on seroma formation (and pre-peritoneal drain output) by 2 techniques in randomised controlled trial.

all male and female patients presented with first occurrence, unilateral inguinal hernia anticipated for laparoscopic TEP are included into study after informed consent. Patients are randomized into "diathermy-preferred" (DP) group and "blunt dissection-preferred" (BDP) group just before commence of operation after general anaethesia. Surgeons are instructed to use monopolar energy as main dissection method for whole operation if possible (DP), where as blunt dissection is the preferred choice in BDP group but it is allowed to use monopolar energy if needed. Total energy time is measured by a specially designed device attaching to the monopolar pedals as accurate as to millisecond (ms). Pre-peritoneal drains are inserted for drainage and removed 23 hours after operation. Energy time, drainage output, ultrasonic seroma sizes at day 1, day 6, 1 month post-operations, recurrence are compared between 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 and below 90
* Male or female patients
* Unilateral inguinal hernia
* First occurrence hernia
* Consent to laparoscopic hernioplasty for inguinal hernia

Exclusion Criteria:

* inguino-scrotal hernia
* Recurrent inguinal hernia
* Incarcerated hernia
* Bilateral inguinal hernia
* Bleeding tendency
* On anti-platelet agent or anti-coagulant
* Significant co-morbidies
* Patients with pacemaker
* Decline or not consent to

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Drain output at 23 hours post-operation | 23 hours post operation
  pre-peritoneal drain output (in ml) at 23 hours post-operation

SECONDARY OUTCOMES:
Seroma at 23 hours post-operation | 23 hours post operation
  Size of seroma at 23 hours post-operation measured by ultrasonography in 3 dimension in mm.
Seroma at 1 week post-operation | 1 week post operation
  Size of seroma at 1 week post-operation measured by ultrasonography in 3 dimension in mm.
Pain score at first week | 1 week
  Pain score at first week (from day 0 to day 6) will be measured in visual analogue scale from 0-10, with 0 is minimum and 10 is maximum score reported by patients.
Seroma at 1 month post-operation | 1 month post-operation
  Size of seroma at 1 month post-operation measured by ultrasonography in 3 dimension in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Joe KM FAN, MS(HKU), Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Surgery, The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan JKM, Liu J, Chen K, Yang X, Xu X, Choi HK, Chan FSY, Chiu KWH, Lo CM. Reply to Comment to: Preperitoneal closed-system suction drainage after totally extraperitoneal hernioplasty in the prevention of early seroma formation: a prospective double-blind randomized controlled trial. Hernia. 2018 Jun;22(3):469-470. doi: 10.1007/s10029-018-1764-6. Epub 2018 Apr 21. No abstract available. PMID 29681018
- [Result] Fan JKM, Liu J, Chen K, Yang X, Xu X, Choi HK, Chan FSY, Chiu KWH, Lo CM. Preperitoneal closed-system suction drainage after totally extraperitoneal hernioplasty in the prevention of early seroma formation: a prospective double-blind randomised controlled trial. Hernia. 2018 Jun;22(3):455-465. doi: 10.1007/s10029-018-1731-2. Epub 2018 Jan 13. PMID 29332240